CLINICAL TRIAL: NCT00336791
Title: Randomized Clinical Trial to Evaluate the Predictive Accuracy of a Gene Expression Profile-Based Test to Select Patients for Preoperative Taxane/Anthracycline Chemotherapy for Stage I-III Breast Cancer
Brief Title: Randomized Clinical Trial to Evaluate the Predictive Accuracy of a Gene Expression for Stage I-II Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0321
Record Dates: First submitted 2006-06-12; First posted 2006-06-14 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Gene Expression; Fluorouracil; Cyclophosphamide; Doxorubicin; Paclitaxel
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorouracil; Cyclophosphamide; Doxorubicin; Paclitaxel; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paclitaxel + Additional FAC/FEC (Experimental): 12 weekly Paclitaxel treatments 80 mg/m^2 by vein (IVPB) over 1 hour + 4 additional FAC or FEC combination chemotherapy treatments; FAC or FEC treatments given once every 3 weeks.
  FAC Chemotherapy: 5-Fluorouracil 500 mg/m^2 intravenous (IV) day 1 & 4 + Doxorubicin 50 mg/m^2 IV day 1 over 72 hour continuous infusion or IV bolus + Cyclophosphamide 500 mg/m^2 IV day 1.
  FEC Chemotherapy: 5-Fluorouracil 500 mg/m^2 IV day 1 + Epirubicin 100 mg/m^2 IV day 1 + Cyclophosphamide 500 mg/m^2 IV day 1.
  Interventions: Drug: 5-Fluorouracil; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Paclitaxel; Drug: Epirubicin
- FAC/FEC (Active Comparator): 6 courses FAC or FEC Combination Chemotherapy
  FAC Chemotherapy: 5-Fluorouracil 500 mg/m^2 intravenous (IV) day 1 & 4 + Doxorubicin 50 mg/m^2 IV day 1 over 72 hour continuous infusion or IV bolus + Cyclophosphamide 500 mg/m^2 IV day 1.
  FEC Chemotherapy: 5-Fluorouracil 500 mg/m^2 IV day 1 + Epirubicin 100 mg/m^2 IV day 1 + Cyclophosphamide 500 mg/m^2 IV day 1.
  Interventions: Drug: 5-Fluorouracil; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Epirubicin

INTERVENTIONS:
Drug: 5-Fluorouracil — FEC Chemotherapy: 500 mg/m^2 IV on day 1 of 21 day cycle.
  FAC Chemotherapy: 500 mg/m^2 IV on day 1 and day 4 of 21 day cycle.
  Other Names: 5-FU; Adrucil; Efudex
Drug: Cyclophosphamide — FAC and FEC Chemotherapy:
  500 mg/m^2 IV on day 1 of 21 day cycle.
  Other Names: Cytoxan; Neosar
Drug: Doxorubicin — FAC Chemotherapy: 50 mg/m^2 IV on day 1 over 72 hour continuous infusion or IV bolus.
  Other Names: AD; Hydroxydaunomycin hydrochloride
Drug: Paclitaxel — 80 mg/m^2 by vein (IVPB) over 1 hour every week for 12 weeks
  Other Names: Taxol
  Arms: Paclitaxel + Additional FAC/FEC
Drug: Epirubicin — FEC: 100 mg/m^2 IV on day 1 of 21 day cycle.

SUMMARY:
Primary Objectives:

1. To prospectively evaluate the predictive accuracy of a previously discovered gene expression profile-based test to foretell pathologic complete response (pCR) to preoperative paclitaxel/FAC (5-fluorouracil, doxorubicin, cyclophosphamide) chemotherapy for stage I-III breast cancer.
2. To evaluate if our genomic predictive test is specific to the paclitaxel/FAC regimen or it also predicts increased sensitivity to FAC only chemotherapy.

Secondary Objectives:

1. To discover a molecular profile that is associated with pCR after FAC chemotherapy alone
2. To establish a prospectively collected gene expression profile data bank of breast cancer for future studies
3. To compare the pCR rates between patients who receive 6 courses FAC and those who receive sequential paclitaxel /FAC chemotherapies.

DETAILED DESCRIPTION:
The new test being studied measures the presence or absence of each of 12,000-15,000 human genes in the cancer using "DNA chip" technology. All of the therapeutic treatment that you will receive is part of the standard of care. Only the biopsy and Deoxyribonucleic acid (DNA) testing is investigational.

Before and during chemotherapy, you will need to have routine clinical and lab tests that are part of your standard of care. These tests may include x-rays such as computed tomography (CT) scan of the liver or lung, bone scan and mammograms, or ultra sonograms of the breast to find out the extent of the cancer at the time of diagnosis. Blood tests (1-2 tablespoon) will be performed before each FAC (5-fluorouracil, doxorubicin, cyclophosphamide) or FEC (5-fluorouracil, epirubicin, cyclophosphamide) chemotherapy end at least once every 2 weeks during weekly paclitaxel therapy to make sure that it is safe to receive further treatment. All of these tests are part of good clinical care and are not considered investigational.

During treatment with FAC or FEC chemotherapy, you will be seen by your physician every 3 weeks. During the weekly paclitaxel treatment you will be seen by your physician every 4-6 weeks. Additional visits may be necessary depending on your clinical course.

During this study, you will be asked to have a fine needle aspiration (FNA) of the cancer in your breast or lymph nodes. The FNA procedure involves insertion of a small needle into the tumor to suction out (aspirate) cells from the cancer 3-4 times in one session. A physician who is trained in this method will perform the procedure. It could be done at the same time when the diagnosis of your cancer is made or it may be done at later time point. The needle aspiration will have to be done before you start any chemotherapy for your cancer. A DNA chip test called transcriptional profiling will be performed on the FNA specimens at M. D. Anderson in Houston (TX, USA). The test will be done to try to predict if an individual is likely to have response to paclitaxel/FAC chemotherapy or not. This study is done to see how accurate this test is. The chemotherapy response prediction test was developed by investigators at Millennium Pharmaceuticals Inc. (Cambridge, MA, USA) and clinical scientists at M. D. Anderson. This research may lead to the development of a commercial diagnostic test.

Only patients who need chemotherapy to improve their chance of cure may participate in this study. Whether you would benefit from chemotherapy or not will be decided by your physician. During this study 18-24 weeks of chemotherapy will be given to you before surgery. It is clear from several large clinical studies that chemotherapy works equally well regardless of whether you receive it before or after breast surgery. By giving chemotherapy before surgery, researchers can study why some cancers respond so well to treatment. You may expect that 80-90% of the time the cancer will shrink and about 15-30% of the time the cancer will completely disappear from the breast or lymph nodes by the time you finish chemotherapy. Many of the patients who experience the complete disappearance of cancer will be cured. The purpose of this research is to find out who these individuals are and develop a test that could identify them at the time of the diagnosis. About 5-10% of patients do not experience any shrinkage of the cancer and may experience growth of the tumor. If the tumor grows during treatment, you will be switched over to another chemotherapy, you may receive radiation treatment, or you may have surgery. What is the best option for you will need to be decided by your treating physician.

You will be randomly assigned (as in the toss of a coin) to one of two treatment groups.

* Participants in the first group will receive weekly treatments with the chemotherapy drug paclitaxel by vein. After completion of 12 paclitaxel treatments, you will receive 4 additional treatments with FAC or FEC combination chemotherapy. The FAC or FEC treatments are given once every 3 weeks. You and your physician will decide together if FAC or FEC is the more appropriate treatment for you. Both of these treatments are believed to be equally effective but FAC is a longer treatment that requires 72-hour infusion whereas FEC can be given in one day. The total length of treatment is 24 weeks after which you will have breast and lymph node surgery.
* Participants in the second group will receive 6 treatments (6 times 3 = 18 weeks) with FAC or FEC before surgery. Those patients who still have cancer in their breast or lymph nodes at the time of surgery may receive additional chemotherapy after the surgery with paclitaxel or a similar drug called docetaxel. One large clinical study showed that addition of 4 courses of paclitaxel after 4 treatments with AC (doxorubicin, cyclophosphamide) chemotherapy improved survival. This is the reason why you may be recommended to receive paclitaxel or docetaxel treatment after surgery. Whether you need additional postoperative chemotherapy or not will need to be discussed between you and your physician.

After you completed all your treatments, you will be contacted (on the phone or by letter) every 6 months for 10 years to find out how well you do and if the cancer has come back.

This research will generate a large database of molecular abnormalities found in breast cancer. Researchers will study the presence or absence of 12,000-15,000 human genes in the cancer of each patient who participates in this study. This information along with the clinical features of the cancer will be stored in the database. The age and race of patients as well as the long-term outcome of treatment will also be included in the database. Other information about your health and family history of cancer may be added to the database in the future. However, your name, address or date of birth will not be part of this research database. The molecular data and the clinical information will be used to learn about the causes of breast cancer and to develop the best individual therapy for future patents.

This is an investigational study. The chemotherapy that you will receive is not experimental. Paclitaxel, FAC or FEC and their combination are commercially available drugs and are all approved by the FDA to treat newly diagnosed breast cancer. A total of up to 273 patients will take part in this multicenter study. Up to 150 may be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed stage I-III invasive carcinoma of the breast for whom adjuvant chemotherapy is indicated. Patients must have intact or measurable residual cancer (by mammogram, ultra sonogram or physical exam) in the breast. Women of childbearing potential must have a negative pregnancy test (serum or urine beta Human chorionic gonadotropin (HCG)) prior to initiation of chemotherapy.
2. Patients should have adequate organ function to tolerate chemotherapy.
3. Patient must be willing to undergo a one-time pretreatment research FNA biopsy

Exclusion Criteria:

1. Patients who have completed lumpectomy, segmental mastectomy or modified radical mastectomy and, therefore no longer have any measurable cancer left in their breast are not eligible.
2. Patients with stage IV, metastatic breast cancers are not eligible.
3. Patients for whom anthracycline or paclitaxel chemotherapies are contraindicated, for example Patients who are pregnant or lactating are not eligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2003-09; Primary Completion 2007-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Pathologic Complete Response Rate in breast and axillary lymph nodes | After completion of preoperative chemotherapy then every 6 months for 10 years.
  Pathologic Complete Response Rate after completion of preoperative chemotherapy, based on routine clinical pathology report where Pathologic complete response defined as complete absence of any viable invasive cancer cells in resected breast and lymph nodes. Specimens in breast may contain in situ cancer (ductal or lobular carcinoma in situ) and still be considered complete response.

CONTACTS AND LOCATIONS:
Overall Officials: Lajos Pusztai, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- UT MD Anderson Cancer Center, Houston, Texas, United States
- Centro Medico Nacional de Occidente, Guadalajara, Mexico
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru
- Grupo Español de Investigacion en Cancer de Mama, Madrid, Spain

REFERENCES:
- [Derived] Desmedt C, Di Leo A, de Azambuja E, Larsimont D, Haibe-Kains B, Selleslags J, Delaloge S, Duhem C, Kains JP, Carly B, Maerevoet M, Vindevoghel A, Rouas G, Lallemand F, Durbecq V, Cardoso F, Salgado R, Rovere R, Bontempi G, Michiels S, Buyse M, Nogaret JM, Qi Y, Symmans F, Pusztai L, D'Hondt V, Piccart-Gebhart M, Sotiriou C. Multifactorial approach to predicting resistance to anthracyclines. J Clin Oncol. 2011 Apr 20;29(12):1578-86. doi: 10.1200/JCO.2010.31.2231. Epub 2011 Mar 21. PMID 21422418
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org